CLINICAL TRIAL: NCT04681547
Title: Ultrasound-guided Genicular Nerve Block: An Analgesic Alternative to LIA for Total Knee Arthroplasty.
Brief Title: Ultrasound-guided Genicular Nerve Block for Total Knee Arthroplasty.
Acronym: PGENECA
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hospital Clinic of Barcelona (Other)
Responsible Party: Principal Investigator, TOMAS MIGUEL CUÑAT LOPEZ, Principal Investigator, Hospital Clinic of Barcelona
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: HCB/2019/1148; 2019-005010-19 (EudraCT Number)
Record Dates: First submitted 2020-12-15; First posted 2020-12-23 (Actual); Last update posted 2021-06-02 (Actual); Status verified 2021-05

CONDITIONS: Pain
Keywords: Pain; Analgesia; LIA; Ultrasound; Genicular Nerve Block
MeSH Terms: conditions — Pain; Agnosia

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Genicular nerve block (Experimental): An ultrasound-assisted genicular nerve block will be performed. 4 ml of 0.2% ropivacaine will be administered, with adrenaline 1: 100 000 in each of the five nerves.
  Interventions: Procedure: Genicular nerve Block
- Local infiltration Analgesia (Active Comparator): Administration of ropivacaine 0.2% 150 ml will be performed.
  Interventions: Procedure: Local Infiltration Analgesia

INTERVENTIONS:
Procedure: Genicular nerve Block — After the administration of spinal anesthesia, the anatomical structures of the proximal and distal region of the knee will be explored through an M- ultrasound machine Turbo® with a high-frequency 6-13 MHz linear probe.
  The ultrasound transducer will be placed in a coronal orientation to the axis of the knee in the corresponding area to be blocked according to anatomical landmarks of superior medial genicular nerve (SMGN), inferior medial genicular nerve block (IMGN), superior lateral genicular nerve (SLGN), inferior lateral genicular nerve (ILGN), and recurrent genicular nerve (RGN).
  It should be noted that the visualization of the genicular arteries in the femoral epicondyles and in the area of the tibial plateau, represents an accurate guide to where the sensory afferents are, however; its display is not constant.
  4 ml of 0.2% ropivacaine will be administered, with adrenaline 1: 100 000 in each of the five nerves.
  Arms: Genicular nerve block
Procedure: Local Infiltration Analgesia — 100 ml of ropivacaine 0.2% with 1 mg of epinephrine during the period of intraoperative ischemia and, before the closure of the surgical wound, 50 ml of ropivacaine 0.2%.
  Arms: Local infiltration Analgesia

SUMMARY:
The hypothesis is to demonstrate the analgesic non-inferiority of the ultrasound-guided geniculate nerve block when compared to the local infiltration analgesia (LIA). It is expected to maintain the quality of analgesia with a selective blockade of the nerves responsible for the sensitive innervation of the knee, reducing the total dose of local anesthetic and adrenaline very markedly.

DETAILED DESCRIPTION:
The main objective is to demonstrate that the ultrasound-guided geniculate nerve block provides not-inferior analgesia to LIA in patients undergoing primary total knee arthroplasty (TKA) in the first 24 hours postoperatively, and during the first mobilization using the numerical evaluation of the pain (NRS).

The secondary objectives are to demonstrate that the consumption of opioids and the range of joint mobility are not inferior in those patients who receive geniculate nerve blocks compared to those who receive LIA.

ELIGIBILITY:
Inclusion Criteria:

* Subjects scheduled for primary elective total knee arthroplasty
* American Society of Anesthesiologists Physical Status I-III
* BMI 18-40 kg/m2

Exclusion Criteria:

* Inability to cooperate with protocol
* Allergy to any medication of protocol
* Contraindication to peripheral nerve block (e.g. local or systemic infection, neurologic deficit or disorder, previous trauma or surgery to ipsilateral knee, etc.)
* Revision or prothesis replacement knee surgery
* Chronic opioid consumption (daily morphine equivalent of >30 mg for at least four weeks prior to surgery)
* Bleeding diathesis or non-pharmacological coagulopathy

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2020-12-15 (Actual); Primary Completion 2021-04-30 (Actual); Study Completion 2021-04-30 (Actual)

PRIMARY OUTCOMES:
NRS at PACU | 1 hour after surgery
  NRS [Numerical Rating Scale, 0-11] at PACU [post-anaesthesia care unit] after spinal block reversal, evaluated as active contralateral knee genuflection at 90 degrees.
NRS at 12 hours after surgery | 12 hours
  Pain will be assessed by NRS [Numerical Rating Scale, 0-11] by a ward nurse, blind for intraoperative analgesic treatment.
NRS at 24 hours after surgery | 24 hours
  Pain will be assessed by NRS [Numerical Rating Scale, 0-11] by a ward nurse, blind for intraoperative analgesic treatment.
NRS after physiotherapy | 24 hours
  It corresponds to day 1 after the surgical intervention and will be carried out in the hospitalization room by a physiotherapist. The NRS [Numerical Rating Scale, 0-11] will be recorded during the first examination and mobilization

SECONDARY OUTCOMES:
Opioid consumption in the postoperative period | until 24 hours
  Opioid consumption in the postoperative period in oral morphine equivalents
Knee mobility range | 24 hours
  Minimal and maximal mobility range [degrees]
Quality of sleep | 24 hours
  Quality of sleep of the first night using the quality of sleep visual analogue scale [0-100 mm]

CONTACTS AND LOCATIONS:
Overall Officials: Tomás López, MD, Principal Investigator — Hospital Clinic of Barcelona; Xavier Sala-Blanch, MD, Principal Investigator — Hospital Clinic of Barcelona
Locations (1):
- Hospital Clínic de Barcelona, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No